CLINICAL TRIAL: NCT02852421
Title: Randomized Prospective Study to Evaluate Efficacy and Safety of Single Versus Multiple Injection Ultrasound Guided Paravertebral Blocks for Breast Surgery
Brief Title: Single Versus Multiple Injection Ultrasound Guided Paravertebral Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Sugantha Ganapathy, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17477
Record Dates: First submitted 2016-07-15; First posted 2016-08-02 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Breast Neoplasms; Anesthesia
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multiple injection paravertebral blocks (Active Comparator): Patients in this group will receive five injections of paravertebral blocks from T1 to T5 level. 5 ml of 0.5% "ropivacaine" was injected at each level.
  Interventions: Procedure: Multiple injection paravertebral blocks
- Single injection paravertebral block (Experimental): Patients in single injection group will receive single injection paravertebral blocks at T3-T4 level with 25 ml of 0.5% "ropivacaine" and four subcutaneous sham injections.
  Interventions: Procedure: Single injection paravertebral block

INTERVENTIONS:
Procedure: Single injection paravertebral block — The patients in single injection group will receive single injection paravertebral block at T3-T4 level with 25 ml of 0.5% "ropivacaine" and four subcutaneous sham injections
  Arms: Single injection paravertebral block
Procedure: Multiple injection paravertebral blocks — Patients in the multiple injection group will receive five injections of paravertebral blocks from T1 to T5 level. 5 ml of 0.5% "ropivacaine" was injected at each level.
  Arms: Multiple injection paravertebral blocks

SUMMARY:
Paravertebral block (PVB) has been shown to provide excellent analgesia for major breast surgeries resulting in reduced narcotic consumption, reduced nausea, improved quality of recovery, reduced chronic pain and possibly reduced metastasis with breast cancer. Traditionally, PVB is done by multiple injections below T1-T5 transverse processes. With multiple injections, the risk is increased for a pleural, an intraneural, and/or an intravascular injection. Recently, ultrasonography is being used to facilitate PVB. The use of ultrasound imaging enables real-time needle visualization during the procedure. This may improve efficacy and reduce the chances of complication like pneumothorax. Currently, there are no data comparing ultrasound-guided single injection technique with multiple injections technique with regards to extent of spread for PVB. Our objective is to investigate the extent of dermatomal spread of PVB when equal volumes of local anesthetic are injected at one versus five paravertebral sites for patients undergoing major breast surgery. In addition, the investigators wish to compare the performance time and duration of analgesia.

Methodology: After local REB approval, 72 patients undergoing a unilateral mastectomy with or without axillary node dissection will be randomized to receive either single or multiple injections PVB. The PVB will be performed in prone position under real-time ultrasound guidance using a para-sagittal approach.The patients in single injection group will receive single injection PVB at T3-T4 level with 25 ml of 0.5% ropivacaine and four subcutaneous sham injections. Patients in the multiple injection group will receive five injections of PVB from T1 to T5 level. 5 ml of 0.5% ropivacaine will be injected at each level. Pleural drift will be used as a sign of correct needle tip location and local anaesthetic spread. The pinprick method will be used to assess the extent of dermatomal blockade, 20 minutes following the completion of procedure. All patients will receive a standardized general anesthesia for the surgery. Any adverse events including pneumothorax, epidural spread, LA toxicity/seizure, total spinal, will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Females, age 18 to 80 years, scheduled to receive unilateral mastectomy surgery, with or without axillary node dissection
* Able to give informed consent
* Able to cooperate with study process
* Availability of home telephone.

Exclusion Criteria:

* Patient refusal or lack of informed consent
* allergy to local anesthetic and other medications used in the study
* Bilateral mastectomies
* Coexisting hematological disorder or with deranged coagulation parameters
* Pre-existing major organ dysfunction such as hepatic and renal failure
* Significant thoracic kyphoscoliosis
* History of previous thoracic surgery.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Sensory dermatomal spread | 20 minutes
  20 minutes after block performance

SECONDARY OUTCOMES:
Time to performance of procedure | Duration of procedure
Cephalic and caudal dermatomal spread | 20 minutes after block performance
Incidence of complication | 24 hours
  Follow-up phone call
VAS pain scores in PACU | 6 hours
  During PACU stay
Duration of self-reported numbness at the surgical site | 24 hours
  At follow-up phone call

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Joseph's Health Care, London, Ontario
  - London Health Sciences Centre University Hospital, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boughey JC, Goravanchi F, Parris RN, Kee SS, Frenzel JC, Hunt KK, Ames FC, Kuerer HM, Lucci A. Improved postoperative pain control using thoracic paravertebral block for breast operations. Breast J. 2009 Sep-Oct;15(5):483-8. doi: 10.1111/j.1524-4741.2009.00763.x. Epub 2009 Jul 13. PMID 19624418
- [Background] Exadaktylos AK, Buggy DJ, Moriarty DC, Mascha E, Sessler DI. Can anesthetic technique for primary breast cancer surgery affect recurrence or metastasis? Anesthesiology. 2006 Oct;105(4):660-4. doi: 10.1097/00000542-200610000-00008. PMID 17006061
- [Background] Cheema S, Richardson J, McGurgan P. Factors affecting the spread of bupivacaine in the adult thoracic paravertebral space. Anaesthesia. 2003 Jul;58(7):684-7. doi: 10.1046/j.1365-2044.2003.03189_1.x. PMID 12886912
- [Background] Lonnqvist PA, MacKenzie J, Soni AK, Conacher ID. Paravertebral blockade. Failure rate and complications. Anaesthesia. 1995 Sep;50(9):813-5. doi: 10.1111/j.1365-2044.1995.tb06148.x. PMID 7573876
- [Background] Naja ZM, El-Rajab M, Al-Tannir MA, Ziade FM, Tayara K, Younes F, Lonnqvist PA. Thoracic paravertebral block: influence of the number of injections. Reg Anesth Pain Med. 2006 May-Jun;31(3):196-201. doi: 10.1016/j.rapm.2005.12.004. PMID 16701182
- [Background] O Riain SC, Donnell BO, Cuffe T, Harmon DC, Fraher JP, Shorten G. Thoracic paravertebral block using real-time ultrasound guidance. Anesth Analg. 2010 Jan 1;110(1):248-51. doi: 10.1213/ANE.0b013e3181c35906. Epub 2009 Nov 21. PMID 19933536
- [Derived] Uppal V, Sondekoppam RV, Sodhi P, Johnston D, Ganapathy S. Single-Injection Versus Multiple-Injection Technique of Ultrasound-Guided Paravertebral Blocks: A Randomized Controlled Study Comparing Dermatomal Spread. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):575-581. doi: 10.1097/AAP.0000000000000631. PMID 28665874